CLINICAL TRIAL: NCT04857671
Title: BACT - Botulinum Toxin A in Frequent and Chronic Tension-type Headache With the FollowTheSutures Paradigm. A Double Blind, Randomized, Placebo-controlled Cross-over Trial
Brief Title: Botulinum Toxin A in Frequent and Chronic Tension-type Headache
Acronym: BACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Norwegian University of Science and Technology (Other); Sandvika Nevrosenter (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 90953; 2019-001385-16 (EudraCT Number)
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Tension-Type Headache
Keywords: Botulinum toxins, type A; Injections
MeSH Terms: conditions — Tension-Type Headache | interventions — Botulinum Toxins, Type A; Saline Waters; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: In this study, injections will follow a slightly modified FollowTheSutures injection protocol.
  Study duration is 36 weeks long. A 4 weeks screening/baseline period with a daily electronic headache diary (eDiary) follows inclusion and informed consent. After completing the 4-week screening/baseline period, participants will be re-screened and eligible participants will enter the randomized phase of the study consisting of two treatment periods. The treatment periods is either injections with verum (onabotulinum toxin suspended in saline (Botox® and NaCl 0,9% Braun) or placebo (only NaCl 0,9% Braun). The participants are randomized to the order with which they enter the two periods, and a quadruple-blinding regime is implemented. Each treatment period lasts 12 weeks, separated by a 4 week washout period. Participants continue to keep a daily eDiary and register adverse events in the entire randomized period.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin A injections (Experimental): Botulinum toxin A (Botox)
  Interventions: Drug: Botulinum Toxin Type A in saline water; Drug: Isotone saline water
- placebo injections (Placebo Comparator): Isotone saline water
  Interventions: Drug: Botulinum Toxin Type A in saline water; Drug: Isotone saline water

INTERVENTIONS:
Drug: Botulinum Toxin Type A in saline water — 100 Allergan units Botulinum toxin A in a total of 2 ml sodium chloride (NaCl) 0,9% Braun.
  5 IU of Botox per injection point (0,1ml); in total 100 IU per 20 injections points.
  Other Names: Botox
Drug: Isotone saline water — 2ml Na Cl (sodium chloride) 0,9% Braun. 0,1ml per injection point in total 20 injections points
  Other Names: Sodium chloride solution; NaCl solution

SUMMARY:
Chronic tension-type headache (CTTH) is an underestimated disabling condition that affects a large number of patients. The treatment options for both episodic tension-type headaches, but especially CTTH are few. Poor long-term effects of existing treatment for CTTH (Sarotex, SSRIs, physiotherapy) are reported. Patients with CTTH also have a high risk of developing drug overdose headache (MOH). Non-drug treatments with physiotherapy or alternative medicine also show poor long-term effects. Literature reviews show that there is surprisingly little research on CTTH. Some small clinical trials report a good effect of treatment with botulinum toxin A, but larger controlled trials are needed to confirm or deny this.

The investigators will study effect of treatment with botulinum toxin A in CTTH in BACT study, and will include participants with both frequent and chronic TTH with 10 or more headache days per month.

If BACT outcomes are positive, this will open a possibility for a new treatment for TTH patients.

DETAILED DESCRIPTION:
BACT studies the efficacy of treatment with botulinum toxin with a follwthestuture injection regime in frequent and chronic tension type headache (TTH). This is be a randomized, placebo-controlled, triple blind, cross-over trial. The primary efficacy variable is the difference in monthly headache days in the active period versus the placebo period. In this study, injections will follow a slightly modified FollowTheSutures injection protocol. Study duration is 36 weeks long. The target population is male and female patients 18 to 75 years of age with TTH, with 10 or more headache days per month.

ELIGIBILITY:
Inclusion criteria:

Eligible participants must meet all of the inclusion criteria in this study.

* Aged 18 to 75 years
* Frequent or chronical tension type headache according to the ICHD-3 (2.2.3) criteria with 10 or more headache days per month
* Headache history of minimum one year.
* Previously unsatisfactory treatment effect, bothersome side-effects to or contra-indications to at least one TTH prophylactic drug.
* Subject agrees to maintain current preventive headache medication regimens (no change in type, frequency, or dose) during the whole study period.
* In case of women of childbearing potential (WOCBP) they have to be using highly effective contraception (for more details below).
* Signed informed consent.

Exclusion criteria

All candidates meeting any of the exclusion criteria at baseline or visit nr.2 will be excluded from study participation:

* Patients with migraine with more than 1 migraine day per month.
* Patients with other forms of primary or secondary headaches; including medication overuse headache (MOH).
* Change in type, dosage or dose frequency of preventive headache medication < 1 months prior to inclusion.
* Previous exposure at any time to any botulinum toxin serotype.
* Pregnancy, breastfeeding or planned pregnancy.
* Patients with diseases that are contraindications for use of BoNT-A (Myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, other diseases interfering with neuromuscular function) or allergy to BoNT-A, or treatment with drugs affecting the neuromuscular junction;
* Active infection at the sites of injection
* Subject has been diagnosed with any major infectious processes such as osteomyelitis, or primary or secondary malignancies involving the face that have been active or required treatment in the past 6 months.
* Any psychiatric disorder that may affect ability to comply with study procedures in the opinion of study investigator.
* Other severe chronical pain conditions.
* Abuse of alcohol or illicit drugs.
* Participating in another trial that might affect the current study.

Contraception for women of childbearing potential (WOCBP) Such methods will include combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence. This group of patients should not be using other drugs that might interact and reduce the efficacy of the used anticonceptive drug. WOCBP is defined as fertile women, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods, include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

Ability to understand study procedures and to comply with them for the entire length of the study. WOCBP will have to agree to take a pregnancy test before the injection with the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Difference in TTH-headache days in week 5-8 of the active period versus the placebo period. | 36 weeks
  Difference in TTH- headache days in week 5-8 of the active period versus the placebo period.

SECONDARY OUTCOMES:
50% responders (50% reduction in TTH-headache days from baseline) in week 1-4, 5-8 and 9-12 | 36 weeks
  50% responders (50% reduction in TTH-headache days from baseline) in week 1-4, 5-8 and 9-12
Difference in TTH-headache days in week 1-4 and 9-12, and in the entire treatment period | 36 weeks
  Difference in TTH-headache days in week 1-4 and 9-12, and in the entire treatment period
30% responders (30% reduction in TTH-headache days from baseline) in week 1-4, 5-8 and 9-12 | 36 weeks
  30% responders (30% reduction in TTH-headache days from baseline) in week 1-4, 5-8 and 9-12
Quality of life score on EQ-5D-5L | 36 weeks
  EQ-5D-5L at week 8 and 12 after injection
Patient Global Impression of Improvement (PGI-I) | 36 weeks
  scale 7-points - (very much better) to 7 (very much worse) 8 and 12 after injection
Average maximum pain intensity in Numeric Rating Scale (NRS from 0 to10) in week 1-4, 5-8 and 9-12 | 36 weeks
  NRS scale: 0 meaning no pain and 10 meaning the worst pain imaginable)
Headache Impact Test (HIT-6) | 36 weeks
  HIT-6 at week 8 and 12 after injection
Average number of headache hours per day in week 1-4, 5-8 and 9-12. | 36 weeks
  Average number of headache hours per day in week 1-4, 5-8 and 9-12.
Average number of days with intake of painkillers per month in week 1-4, 5-8 and 9-12 | 36 weeks
  Average number of days with intake of painkillers per month in week 1-4, 5-8 and 9-12
Acceptability | 36 weeks
  Acceptability
Difference in occurrence of adverse events and serious adverse events in the active period and the placebo period | 36 weeks
  Difference in occurrence of adverse events and serious adverse events in the active period and the placebo period

OTHER OUTCOMES:
e the efficacy of BoNT in treatment group as compared to placebo group in reducing the area-under-the-headache curve (AUC) | recorded daily as ePROMs in an eDiary throughout the study participation.
  Tertiary/Exploratory objective and endpoints Exploratory objective: To investigate the efficacy of BoNT in treatment group as compared to placebo group in reducing the area-under-the-headache curve (AUC). This variable defined according to IHS-guidelines(22) Exploratory endpoint: To investigate the efficacy of BoNT in treatment group as compared to placebo group in reducing the area-under-the-headache curve (AUC).
  The area-under-the-headache curve (AUC) is validated and recommended by the International Headache Society for controlled trials of preventive treatment of TTH in adults . The AUC measurement combines headache intensity and headache duration, and it will provide more insights to how the burden of headache has changed after the intervention than the primary efficacy measures (days with TTH).
  AUC is defined accordingly as the sum of the daily recordings of the headache duration multiplied with the headache intensity (also called headache index).

CONTACTS AND LOCATIONS:
Overall Officials: Norunn Hanssen Hestvik, Study Director — Clinic for Medicine and rehabilitation, Nord Trøndelag Trust HNT
Locations (1):
- Namsos Sykehus, Namsos, Norway

IPD SHARING:
Plan to Share IPD: No